CLINICAL TRIAL: NCT02378935
Title: A Phase 2, Global, Multicenter, Open-Label Study to Investigate the Safety and Efficacy of GS-9857 Plus Sofosbuvir/GS-5816 Fixed Dose Combination in Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Safety and Efficacy of Voxilaprevir Plus Sofosbuvir/Velpatasvir Fixed Dose Combination in Adults With Chronic Genotype 1 HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-1168
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — voxilaprevir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- VOX+SOF/VEL 6 wk, TN, without cirrhosis (Experimental): VOX + SOF/VEL for 6 weeks (treatment naive (TN), without cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL 8 wk, TN, without cirrhosis (Experimental): VOX + SOF/VEL for 8 weeks (treatment naive, without cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL 6 wk, TN, with cirrhosis (Experimental): VOX + SOF/VEL for 6 weeks (treatment naive, with cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL 8 wk, TN, with cirrhosis (Experimental): VOX + SOF/VEL for 8 weeks (treatment naive, with cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL+RBV 8 wk, TN, with cirrhosis (Experimental): VOX + SOF/VEL+RBV for 8 weeks (treatment naive, with cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL; Drug: RBV
- VOX+SOF/VEL 8 wk, DAA-E, without cirrhosis (Experimental): VOX + SOF/VEL for 8 weeks (direct-acting antiviral experienced (DAA-E), without cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL 12 wk, DAA-E, without cirrhosis (Experimental): VOX + SOF/VEL for 12 weeks (direct-acting antiviral experienced, without cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL 8 wk, DAA-E, with cirrhosis (Experimental): GS-9857 + SOF/VEL for 8 weeks (direct-acting antiviral experienced, with cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL 12 wk, DAA-E, with cirrhosis (Experimental): GS-9857 + SOF/VEL for 12 weeks (direct-acting antiviral experienced, with cirrhosis)
  Interventions: Drug: VOX; Drug: SOF/VEL
- VOX+SOF/VEL 12 wk (GS-US-338-1121) (Experimental): VOX + SOF/VEL for 12 weeks (participants who were previously enrolled in GS-US-338-1121 phase 1b study)
  Interventions: Drug: VOX; Drug: SOF/VEL

INTERVENTIONS:
Drug: VOX — 100 mg tablet(s) administered orally once daily with food
  Other Names: GS-9857
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily with food
  Other Names: GS-7977/GS-5816; Epclusa®
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: VOX+SOF/VEL+RBV 8 wk, TN, with cirrhosis

SUMMARY:
This primary objectives of the study are to evaluate the safety, tolerability, and efficacy of voxilaprevir (VOX) plus sofosbuvir/velpatasvir (SOF/VEL) fixed dose combination (FDC) ± ribavirin (RBV) in adults with chronic genotype 1 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with chronic HCV infection
* HCV RNA ≥10^4 IU/mL at screening
* HCV genotype 1
* Cirrhosis determination; a liver biopsy may be required
* Screening laboratory values within defined thresholds
* Use of two contraception methods if female of childbearing potential or sexually active male

Key Exclusion Criteria:

* Pregnant or nursing female
* Current or prior history of hepatic decompensation
* Hepatocellular carcinoma (HCC) or other clinically significant malignancy
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment or compliance with the protocol

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (34):
- United States (31):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Huntington Memorial Hospital Liver Center, Pasadena, California
  - Medical Associates Research Group, Inc., San Diego, California
  - University of Colorado, Denver, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Orlando Immunology center, Orlando, Florida
  - South Florida Center of Gastroenterology, P.A., Wellington, Florida
  - Center for Hep C/Atlanta Medical Center, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Indianapolis Gastroenterology & Hepatology, Inc., Indianapolis, Indiana
  - Beth Isreal Deconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital and Health System, Detroit, Michigan
  - ID Care, Hillsborough, New Jersey
  - Southwest Care Center, Santa Fe, New Mexico
  - North Shore/Long Island Jewish PRIME, Manhasset, New York
  - Mount Sinai Beth Israel, New York, New York
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - UPMC Center for Liver Diseases, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastro One, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Inc., Nashville, Tennessee
  - Texas Liver Institute, San Antonio, Texas
  - Liver Institute of Virginia, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clinical Studies Trust, Christchurch
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Lawitz E, Reau N, Hinestrosa F, Rabinovitz M, Schiff E, Sheikh A, Younes Z, Herring R Jr, Reddy KR, Tran T, Bennett M, Nahass R, Yang JC, Lu S, Dvory-Sobol H, Stamm LM, Brainard DM, McHutchison JG, Pearlman B, Shiffman M, Hawkins T, Curry M, Jacobson I. Efficacy of Sofosbuvir, Velpatasvir, and GS-9857 in Patients With Genotype 1 Hepatitis C Virus Infection in an Open-Label, Phase 2 Trial. Gastroenterology. 2016 Nov;151(5):893-901.e1. doi: 10.1053/j.gastro.2016.07.039. Epub 2016 Jul 30. PMID 27486034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States and New Zealand. The first participant was screened on 17 February 2015. The last study visit occurred on 12 April 2016.
Pre-assignment Details: 255 participants were screened. Enrollment was sequential, with the longer treatment duration groups enrolled, treated, and evaluated for Sustained Virologic Response 4 Weeks After Discontinuation of Therapy (SVR4) prior to enrollment of the shorter treatment duration groups, which were not enrolled, at the discretion of the Sponsor.
Groups:
- VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic: Voxilaprevir (VOX) 100 mg tablet + sofosbuvir/veltapasvir (Epclusa® ; SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet administered once daily for 6 weeks in treatment naive participants without cirrhosis
- VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet administered once daily for 8 weeks in treatment naive participants without cirrhosis
- VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet administered once daily for 8 weeks in treatment naive participants with cirrhosis
- VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) administered once daily for 8 weeks in treatment naive participants with cirrhosis
- VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet administered once daily for 12 weeks in direct-acting antiviral (DAA) experienced participants without cirrhosis
- VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet administered once daily for 12 weeks in DAA-experienced participants with cirrhosis
- VOX+SOF/VEL 12 Weeks (GS-US-338-1121): VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet administered once daily for 12 weeks in participants who were previously enrolled in Gilead sponsored phase 1b study GS-US-338-1121
Period: Overall Study
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
Started | 34 | 36 | 33 | 31 | 31 | 32 | 8
Completed | 24 | 36 | 30 | 25 | 31 | 32 | 8
Not Completed | 10 | 0 | 3 | 6 | 0 | 0 | 0
Not completed — Lack of Efficacy | 10 | 0 | 2 | 6 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet administered once daily for 6 weeks in treatment naive participants without cirrhosis
- VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC administered once daily for 8 weeks in treatment naive participants without cirrhosis
- VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet + RBV tablets (1000 or 1200 mg daily based on weight) administered once daily for 8 weeks in treatment naive participants with cirrhosis
- VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic: VOX 100 mg tablet + SOF/VEL (400/100 mg) FDC tablet administered once daily for 12 weeks in DAA-experienced participants without cirrhosis
- Total: Total of all reporting groups
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121) | Total
Number analyzed (Participants) | 34 | 36 | 33 | 31 | 31 | 32 | 8 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.5) | 51 (14.3) | 58 (7.2) | 59 (6.7) | 57 (7.8) | 59 (6.5) | 5.7 (5.9) | 56 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 14 | 12 | 8 | 6 | 5 | 71
  Male | 23 | 21 | 19 | 19 | 23 | 26 | 3 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 4 | 7 | 5 | 4 | 6 | 0 | 29
  White | 31 | 32 | 25 | 26 | 27 | 26 | 8 | 175
  Native Hawaiian or Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8 | 7 | 4 | 10 | 5 | 42
  Not Hispanic or Latino | 31 | 31 | 25 | 24 | 27 | 22 | 3 | 163
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 36 | 28 | 31 | 31 | 32 | 8 | 198
  New Zealand | 2 | 0 | 5 | 0 | 0 | 0 | 0 | 7
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 12 | 9 | 7 | 12 | 4 | 4 | 3 | 51
    CT | 15 | 21 | 19 | 12 | 19 | 21 | 3 | 110
    TT | 7 | 4 | 7 | 6 | 7 | 7 | 2 | 40
    Missing | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 4
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.51) | 6.2 (0.55) | 6.0 (0.59) | 6.3 (0.47) | 6.4 (0.77) | 6.0 (0.61) | 6.5 (0.38) | 6.2 (0.60)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 6 | 10 | 14 | 6 | 6 | 16 | 0 | 58
  ≥ 800,000 IU/mL | 28 | 26 | 19 | 25 | 25 | 16 | 8 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set (FAS): participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
Number analyzed (Participants) | 34 | 36 | 33 | 31 | 31 | 32 | 8
percentage of participants | 70.6 [52.5 to 84.9] | 100.0 [90.3 to 100.0] | 93.9 [79.8 to 99.3] | 80.6 [62.5 to 92.5] | 100 [88.8 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [63.1 to 100.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 Weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
Number analyzed (Participants) | 34 | 36 | 33 | 31 | 31 | 32 | 8
percentage of participants | 0 | 0 | 0 | 6.5 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
Number analyzed (Participants) | 34 | 36 | 33 | 31 | 31 | 32 | 8
percentage of participants
  SVR4 | 88.2 [72.5 to 96.7] | 100.0 [90.3 to 100.0] | 93.9 [79.8 to 99.3] | 87.1 [70.2 to 96.4] | 100.0 [88.8 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [63.1 to 100.0]
  SVR24 | 70.6 [52.5 to 84.9] | 100.0 [90.3 to 100.0] | 93.9 [79.8 to 99.3] | 80.6 [62.5 to 92.5] | 100.0 [88.0 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [63.1 to 100.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Baseline through end of treatment (Week 6, Week 8 or Week 12, as applicable)
Population: Participants in the Full Analysis Set with available data were analyzed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
Number analyzed (Participants) | 34 | 36 | 33 | 31 | 31 | 32 | 8
percentage of participants
  Week 1 | 23.5 [10.7 to 41.2] | 38.9 [23.1 to 56.5] | 33.3 [18.0 to 51.8] | 16.1 [5.5 to 33.7] | 22.6 [9.6 to 41.1] | 28.1 [13.7 to 46.7] | 12.5 [0.3 to 52.7]
  Week 2 | 79.4 [62.1 to 91.3] | 75.0 [57.8 to 87.9] | 63.6 [45.1 to 79.6] | 54.8 [36.0 to 72.7] | 58.1 [39.1 to 75.5] | 62.5 [43.7 to 78.9] | 75.0 [34.9 to 96.8]
  Week 4 | 100.0 [89.7 to 100.0] | 94.4 [81.3 to 99.3] | 90.9 [75.7 to 98.1] | 96.8 [83.3 to 99.9] | 93.5 [78.6 to 99.2] | 96.9 [83.8 to 99.9] | 100.0 [63.1 to 100.0]
  Week 6: number analyzed (Participants) | 34 | 36 | 33 | 30 | 31 | 32 | 8
  Week 6 | 100.0 [89.7 to 100.0] | 100.0 [90.3 to 100.0] | 97.0 [84.2 to 99.9] | 100.0 [88.4 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [63.1 to 100.0]
  Week 8: number analyzed (Participants) | 0 | 36 | 33 | 31 | 31 | 32 | 8
  Week 8 |  | 100.0 [90.3 to 100.0] | 100.0 [89.4 to 100.0] | 100.0 [88.4 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [63.1 to 100.0]
  Week 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 31 | 32 | 8
  Week 10 |  |  |  |  | 100.0 [88.8 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [63.1 to 100.0]
  Week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 31 | 32 | 8
  Week 12 |  |  |  |  | 100.0 [88.8 to 100.0] | 100.0 [89.1 to 100.0] | 100.0 [63.1 to 100.0]

5. Secondary Outcome: HCV RNA Change From Baseline
Time Frame: Baseline through end of treatment (Week 6, Week 8 or Week 12, as applicable)
Population: Participants in the Full Analysis Set with available data were analyzed
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
Number analyzed (Participants) | 34 | 36 | 33 | 31 | 31 | 32 | 8
log10 IU/mL
  Change at Week 1 | -4.64 (0.556) | -4.60 (0.595) | -4.15 (0.733) | -4.31 (0.658) | -4.40 (0.577) | -4.19 (0.504) | -4.71 (0.486)
  Change at Week 2 | -5.00 (0.504) | -4.98 (0.519) | -4.57 (0.662) | -4.85 (0.583) | -4.97 (0.711) | -4.66 (0.520) | -5.27 (0.450)
  Change at Week 4: number analyzed (Participants) | 34 | 36 | 33 | 30 | 31 | 32 | 8
  Change at Week 4 | -5.07 (0.514) | -5.06 (0.534) | -4.81 (0.576) | -5.17 (0.481) | -5.22 (0.755) | -4.84 (0.601) | -5.35 (0.385)
  Change at Week 6: number analyzed (Participants) | 34 | 36 | 33 | 30 | 31 | 32 | 8
  Change at Week 6 | -5.07 (0.514) | -5.08 (0.549) | -4.84 (0.586) | -5.16 (0.480) | -5.24 (0.767) | -4.84 (0.611) | -5.35 (0.385)
  Change at Week 8: number analyzed (Participants) | 0 | 36 | 33 | 30 | 31 | 32 | 8
  Change at Week 8 |  | -5.08 (0.549) | -4.85 (0.591) | -5.16 (0.480) | -5.24 (0.767) | -4.84 (0.611) | -5.35 (0.385)
  Change at Week 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 31 | 32 | 8
  Change at Week 10 |  |  |  |  | -5.24 (0.767) | -4.84 (0.611) | -5.35 (0.385)
  Change at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 31 | 32 | 8
  Change at Week 12 |  |  |  |  | -5.24 (0.767) | -4.84 (0.611) | -5.35 (0.385)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
Number analyzed (Participants) | 34 | 36 | 33 | 31 | 31 | 32 | 8
percentage of participants | 29.4 | 0 | 6.1 | 19.4 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic | VOX+SOF/VEL 12 Weeks (GS-US-338-1121)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36 | 0/33 | 0/31 | 0/31 | 0/32 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36 | 2/33 | 0/31 | 0/31 | 0/32 | 0/8
Other Adverse Events (participants affected / at risk) | 21/34 | 20/36 | 18/33 | 24/31 | 15/31 | 16/32 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic (N=34) | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic (N=36) | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic (N=33) | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic (N=31) | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic (N=31) | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic (N=32) | VOX+SOF/VEL 12 Weeks (GS-US-338-1121) (N=8)
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VOX+SOF/VEL 6 Weeks, Treatment Naive, Non Cirrhotic (N=34) | VOX+SOF/VEL 8 Weeks, Treatment Naive, Non Cirrhotic (N=36) | VOX+SOF/VEL 8 Weeks, Treatment Naive, Cirrhotic (N=33) | VOX+SOF/VEL+RBV 8 Weeks, Treatment Naive, Cirrhotic (N=31) | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Non Cirrhotic (N=31) | VOX+SOF/VEL 12 Weeks, DAA-Experienced, Cirrhotic (N=32) | VOX+SOF/VEL 12 Weeks (GS-US-338-1121) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 3 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 6 | 2 | 3 | 3 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 10 | 7 | 9 | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 7 | 1 | 10 | 7 | 3 | 2
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 11 | 7 | 7 | 9 | 4 | 5 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 5 | 1 | 0 | 3 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years